CLINICAL TRIAL: NCT00195156
Title: Phase I Trial of ATRA-IV and Depakote in Patients With Advanced Solid Tumor Malignancies
Brief Title: Treatment With ATRA-IV and Depakote in Patients With Advanced Solid Tumor Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1002-536
Record Dates: First submitted 2005-09-14; First posted 2005-09-19 (Estimated); Last update posted 2006-09-14 (Estimated); Status verified 2006-09

CONDITIONS: Solid Tumor Malignancies
Keywords: Solid Tumor Malignancies
MeSH Terms: interventions — Valproic Acid

INTERVENTIONS:
Drug: ATRA-IV
Drug: Depakote

SUMMARY:
The purpose of this study is to find out the highest tolerated dose of Depakote in combination with liposome encapsulated all-trans retinoic acid (ATRA-IV) in patients with advanced solid tumor malignancies.

DETAILED DESCRIPTION:
To determine the maximum tolerated dose of Depakote in combination with liposome encapsulated all-trans retinoic acid (ATRA-IV) in patients with advanced solid tumor malignancies.

This will be a 2-step dose escalation study. Once the patient starts therapy at a designated dose level, it will not be escalated for that patient. Three patients at each dose level must complete 4 weeks of therapy before escalating to the next higher level. If none of the patients experience dose limiting toxicity (DLT), then 3 new patients will be treated with the next higher dose level.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologic confirmation of a solid tumor malignancy with clinical evidence of metastatic disease.
* Patients must have failed at least one standard therapy, if available, for their malignancy. Patients may be entered on the trial without prior therapy if there is no standard effective therapy available.
* No active brain metastases or epidural tumor.

Exclusion Criteria:

* Concomitant administration of steroids.
* Irradiation or chemotherapy within 14 days of start of protocol.
* Evidence of another active cancer, except for non-melanoma, carcinoma of the skin and in-situ carcinoma of the cervix curatively treated, Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for greater than 5 years.
* Women who are pregnant or lactating. Women or men of reproductive age who are unwilling to use two forms of effective contraception.
* Patients with clinically significant cardiac, renal or hepatic disease; severe debilitating pulmonary disease; or history of diabetes mellitus prone to ketoacidosis.
* Patients with a history of pancreatitis.
* Patients with known hypersensitivity to retinoids or retinoic acid derivatives.
* Patients with coagulation disorders, such as thrombophlebitis or pulmonary embolism.
* Patients with pre-existing psychiatric condition, especially depression or a history of severe uncontrolled psychiatric disorder.
* Patients with pre-existing thyroid abnormalities whose thyroid function cannot be maintained in the normal range.
* Patients with chronic moderate to severe nausea.
* Patients with history of epilepsy or a seizure disorder taking anti-convulsant medication.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-07

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of Depakote in combination with liposome encapsulated all-trans retinoic acid (ATRA-IV) in patients with advanced solid tumor malignancies.
To define the dose limiting and other toxicities of the combination therapy
To determine the dosing that should be used in future safety and efficacy (Phase II) trials

SECONDARY OUTCOMES:
To study retinoic acid receptor expression and histone acetylation status to ascertain biologic effect on peripheral blood mononuclear cells and tissue obtained from selected patients who undergo tumor biopsies.
To assess for tumor responses to combination therapy.

CONTACTS AND LOCATIONS:
Overall Officials: David Nanus, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States

REFERENCES:
- [Derived] Orfali N, O'Donovan TR, Cahill MR, Benjamin D, Nanus DM, McKenna SL, Gudas LJ, Mongan NP. All-trans retinoic acid (ATRA)-induced TFEB expression is required for myeloid differentiation in acute promyelocytic leukemia (APL). Eur J Haematol. 2020 Mar;104(3):236-250. doi: 10.1111/ejh.13367. Epub 2020 Jan 13. PMID 31811682